CLINICAL TRIAL: NCT02142725
Title: Randomized, Double-blind, Double-dummy, Placebo-controlled, Phase III Clinical Trial on the Efficacy and Safety of a 12-weeks add-on Treatment With LT 02 vs. Placebo in Patients With Ulcerative Colitis Refractory to Standard Treatment With Mesalamine
Brief Title: Phosphatidylcholine (LT-02) for Induction of Remission in Ulcerative Colitis
Acronym: PROTECT-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: IDMC recommendation
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCG-2/UCA; 2012-003702-27 (EudraCT Number)
Record Dates: First submitted 2014-05-15; First posted 2014-05-20 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LT-02 (Experimental): LT-02 0.8g four times daily
  Interventions: Drug: LT-02
- B: LT-02 (Experimental): LT-02 1.6g twice daily
  Interventions: Drug: LT-02
- Placebo (Placebo Comparator): LT-02 Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LT-02 — four times per day
  Arms: LT-02
Drug: LT-02 — two times per day
  Arms: B: LT-02
Drug: Placebo — four times per day
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare two different dosing regimens of phosphatidylcholine versus placebo for the induction of remission in ulcerative colitis patients non-responsive to standard mesalamine treatment.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of ulcerative colitis
* Active ulcerative colitis disease extent ≥ 15 cm
* Active disease despite treatment with mesalamine

Exclusion Criteria:

* Crohn's disease, indeterminate colitis, ischemic colitis, radiation colitis, microscopic colitis, diverticular disease associated colitis,
* Toxic megacolon or fulminant colitis
* Colon resection
* Evidence of infectious colitis
* Celiac disease
* Bleeding hemorrhoids
* History or presence of ischemic heart disease, myocardial infarction, peripheral arterial disease, ischemic stroke, or transient ischemic attack
* Any severe concomitant renal, endocrine, or psychiatric disorder
* Any relevant known systemic disease
* History of cancer in the last five years
* Abnormal hepatic function or liver cirrhosis
* Abnormal HbA1c at screening visit
* Patients with known hypersensitivity to soy
* Known intolerance/hypersensitivity to Investigational Medicinal Product (IMP)
* Treatment with steroids/methotrexate/Tumor necrosis factor-alpha-antagonists/azathioprine/ 6-mercaptopurine/anti-integrin/coumarins
* Treatment with other investigational drug
* Existing or intended pregnancy or breast-feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2014-07-21 (Actual); Primary Completion 2016-11-11 (Actual); Study Completion 2016-12-16 (Actual)

PRIMARY OUTCOMES:
Rate of clinical remission | 12 weeks

SECONDARY OUTCOMES:
Rate of patients with clinical improvement | 12 weeks
Time to first resolution of symptoms | 12 weeks
Number of stools per week | 12 weeks
Number of days with urgency per week | 12 weeks
Rate of mucosal healing | 12 weeks
Rate of histologic remission | 12 weeks
Physician's global assessment at final visit | 12 weeks
Quality of life | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Axel Dignass, MD, Principal Investigator — Agaplesion Markus-Krankenhaus, 1st Dept. of Medicine
Locations (1):
- Agaplesion Markus-Krankenhaus, 1st Dept. of Medicine, Frankfurt a.M., Germany

REFERENCES:
- [Derived] Dignass A, Stremmel W, Horynski M, Poyda O, Armerding P, Fellermann K, Langhorst J, Kuehbacher T, Uebel P, Stein J, Novacek G, Avalueva E, Oliinyk O, Hasselblatt P, Dorofeyev A, Heinemann H, Mueller R, Greinwald R, Reinisch W; International PROTECT-1/2 Study Groups. Modified-Release Phosphatidylcholine (LT-02) for Ulcerative Colitis: Two Double-Blind, Randomized, Placebo-Controlled Trials. Clin Gastroenterol Hepatol. 2024 Apr;22(4):810-820.e7. doi: 10.1016/j.cgh.2023.09.031. Epub 2023 Oct 6. PMID 37806372